CLINICAL TRIAL: NCT04175626
Title: BIOTRONIK - A Prospective Multicenter Study to Confirm the SaFety and Effectiveness of the Orsiro SiroLimus Eluting Coronary Stent System in the Treatment Of Subjects With up to Three De Novo or Restenotic Coronary Artery Lesions - VII
Brief Title: Safety and Effectiveness of the Orsiro Sirolimus Eluting Coronary Stent System in Subjects With Coronary Artery Lesions
Acronym: BIOFLOW-VII
Status: Active, not recruiting | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIOFLOW-VII
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease; Atherosclerosis, Coronary; Myocardial Ischemia; Ischemic Heart Disease; Acute Coronary Syndrome; Angina Pectoris
Keywords: Drug eluting coronary stents; Sirolimus; Bioabsorbable polymer; DES
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Orsiro sirolimus coronary stent system: Intervention with a Orsiro DES.
  Interventions: Device: Orsiro DES

INTERVENTIONS:
Device: Orsiro DES — Orsiro is a device/drug combination product composed of two components, a device (coronary stent system including a cobalt chromium stent platform), and a drug product (a formulation of sirolimus) contained in a bioabsorbable polymer coating.
  Other Names: Orsiro sirolimus coronary stent system

SUMMARY:
The objective of this post-approval study is to confirm that the clinical performance of the Orsiro stent in a real-world setting is similar to the clinical performance observed for Orsiro in the BIOFLOW-V Investigational Device Exemption pivotal trial, as a condition of the US Food and Drug Administration (FDA) approval (P170030).

DETAILED DESCRIPTION:
BIOFLOW-VII is a prospective, multicenter, single-arm study. Subjects with coronary artery disease (CAD) who undergo an on-label percutaneous coronary intervention (PCI) with a placed Orsiro stent within the prior 24 hours will be screened post-index procedure per the protocol inclusion and exclusion criteria.

Following the index procedure and study enrollment, subjects will be followed for 5 years. The follow-up schedule will include an intermediate study visit at 1 month, a primary endpoint study visit at 12 months, and long-term study visits at 2, 3, 4, and 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age.
2. Subject was an acceptable candidate for treatment with a drug eluting stent at the qualifying index procedure, in accordance with the applicable guidelines on percutaneous coronary interventions and manufacturer's Instructions for Use.
3. Subject received at least one Orsiro stent during an index procedure occurring within 24 hours prior to informed consent, as assessed by the end time of procedure. If more than one stent was implanted during the index procedure, all stents were Orsiro stents.
4. Subject is eligible for dual antiplatelet therapy (DAPT) treatment with aspirin plus either clopidogrel, prasugrel, ticagrelor or ticlopidine.
5. Subject is willing to comply with study follow-up requirements.
6. Subject has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site. Legally authorized representatives are not allowed to consent on a subject's behalf.

Each target lesion/vessel must have met all of the following angiographic criteria from the index procedure for the subject to be eligible for the trial:

1. Subject has up to three target lesions in up to two separate target vessels (two target lesions in one vessel and one target lesion in a separate vessel).
2. Target lesion must be de novo or restenotic lesion in native coronary artery; restenotic lesion must have been treated with a standard PTCA only.
3. Target lesion must be in major coronary artery or branch (target vessel).
4. Target lesion must have angiographic evidence of ≥ 50% and < 100% stenosis (by operator visual estimate). If the target lesion is < 70% stenosed, there should be clinical evidence of ischemia.
5. Target vessel must have a Thrombolysis In Myocardial Infarction (TIMI) flow > 1.
6. Target lesion must be ≤ 36 mm in length by operator visual estimate.
7. Target vessel must have a reference vessel diameter of 2.25-4.0 mm by operator visual estimate.
8. Target lesion must have been treated with a maximum of two overlapping stents.

Exclusion Criteria:

1. Subject had clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation MI (STEMI) within 72 hours prior to the index procedure.
2. Subject is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study.
3. Subject has a known allergy to contrast medium that cannot be adequately pre-medicated, or any known allergy to thienopyridine, aspirin, both heparin and bivalirudin, L-605 cobalt-chromium (Co-Cr) alloy or one of its major elements (cobalt, chromium, tungsten and nickel), silicon carbide, PLLA, sirolimus.
4. Revascularization of any target vessel within 9 months prior to the index procedure or previous PCI of any non-target vessel within 30 days prior to the index procedure or any PCI planned within the next 1 year.
5. Presence of an untreated clinically significant stenosis post-procedure whether treatment is planned or not.
6. Planned surgery within 6 months of index procedure unless DAPT can be maintained throughout the peri-surgical period.
7. History of a stroke or transient ischemic attack (TIA) within 6 months prior to the index procedure.
8. Subject has documented LVEF < 30% prior to consent.
9. Subject is dialysis-dependent.
10. Subject has impaired renal function (blood creatinine > 2.5 mg/dL or 221 μmol/L prior to the index procedure).
11. Subject has leukopenia (i.e. < 3,000 white blood cells/mm3), thrombocytopenia (i.e. < 100,000 platelets/mm3) or thrombocytosis (i.e. > 700,000 platelet/mm3).
12. Any significant concurrent medical diagnosis that would potentially impact DAPT effectiveness or increase thrombotic risk.
13. Subject is receiving chronic anticoagulation (e.g. coumadin, dabigatran, apixaban, rivaroxaban or any other agent).
14. Subject has life expectancy of < 1 year.
15. Subject is participating in an investigational (medical device or drug) clinical study. Subjects may be concurrently enrolled in a post-market study, as long as the post-market study device, drug or protocol does not interfere with the follow-up requirements of this study or does not involve a drug that may confound the interpretation of any relevant clinical events of interest (e.g. investigational DAPT therapy).
16. In the investigator's opinion, subject will not be able to comply with the follow-up requirements.

Subjects will be excluded from the trial if any of the target lesions/vessels met any of the following angiographic criteria during the index procedure:

1. Target lesion was located within or treated through a saphenous vein graft or arterial graft.
2. Target lesion was a restenotic lesion that was previously treated with a bare metal or drug-eluting stent (in-stent restenosis).
3. Target lesion had any of the following characteristics:

   1. Lesion location is within the left main coronary artery, or within 3 mm of the origin of the left anterior descending (LAD) or left circumflex (LCX).
   2. Involves a side branch of > 2.0 mm in diameter.
4. Target vessel/lesion was excessively tortuous/angulated or is severely calcified, that would prevent complete inflation of an angioplasty balloon. This assessment should be based on visual estimation.
5. Target vessel had angiographic evidence of thrombus.
6. Target lesion was totally occluded (100% stenosis).
7. Target vessel was treated with brachytherapy any time prior to the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease (CAD), including those with diabetes mellitus, with symptomatic heart disease, stable angina, unstable angina, non-ST elevation myocardial infarction or documented silent ischemia due to atherosclerotic lesions in the native coronary arteries with a reference vessel diameter of 2.25 mm to 4.0 mm and a lesion length of ≤ 36 mm.
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute
Locations (33):
- United States (33):
  - Cardiology Associates of Mobile, Fairhope, Alabama
  - John Muir Medical Center, Concord, California
  - St. Joseph Hospital Orange, Orange, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Tampa, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Ascension St. Vincent Medical Group, Indianapolis, Indiana
  - Ascension Via Christi Hospitals, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Northern Light Cardiology, Bangor, Maine
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Saint Michael's Medical Center, Newark, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Mercy Health - St Vincent Medical Center, Toledo, Ohio
  - Penn State Health Holy Spirit Medical Center, Camp Hill, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seton Medical Center Austin, Austin, Texas
  - Austin Heart, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - UT Health Science Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Charleston Area Medical Center Memorial Hospital, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Applicable de-identified individual participant data will be made available to achieve aims in approved proposals, including but not limited to sub-analysis or meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning no later than 12 months and ending no earlier than 3 years following initial publication of clinical study results.
Access Criteria: Researchers who provide a methodologically sound proposal for analysis that is not pre-planned or already approved with another researcher. Proposals must be approved by BIOTRONIK and Study Principal Investigator.
  Proposals should be directed to BIOTRONIK Clinical Studies (BIOTRONIK Inc., Attn: Clinical Studies, 6024 Jean Road, Lake Oswego, OR 97035; 1-800-547-0394). To gain access, data requesters will need to sign a data use/access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Orsiro Sirolimus Coronary Stent System
Started | 556
Completed (All subjects included in analysis through 360 days post index procedure.) | 531
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193
  Male | 363
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 513
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 51
  White | 452
  More than one race | 0
  Unknown or Not Reported | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Target Lesion Failure (TLF) at 12 Months Post-Index Procedure
Description: TLF is defined as all cardiac death, target vessel Q-wave or non-Q-wave myocardial infarction (MI), or clinically driven target lesion revascularization (TLR).
Time Frame: 12-Months
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 531
Participants | 9
Statistical Analysis 1: Comparison: Orsiro Sirolimus Coronary Stent System; The primary endpoint was evaluated by performing an exact, binomial test comparing the rate of TLF for the Orsiro stent at 1 year to a performance goal of 6.9%, with Type I error (alpha) of 0.025 and power of 80%. The null hypothesis (Ho) was stated as: The TLF rate of the Orsiro stent at 1 year is greater than or equal to 6.9%. The alternative hypothesis (Ha) was stated as: The TLF rate of the Orsiro stent at 1 year is less than 6.9%; Test type: Superiority; p < 0.0001, Exact, binomial

2. Secondary Outcome: All-cause Death
Time Frame: at Hospital Discharge an average of 1 day, at 1 Month, at 1 Year
Population: Analysis population for each outcome measure time frame is based on participants completing or experiencing an event at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants
  Hospital Discharge | 1
  1 Month: number analyzed (Participants) | 554
  1 Month | 2
  1 Year: number analyzed (Participants) | 536
  1 Year | 6

3. Secondary Outcome: Protocol-defined Any-vessel Myocardial Infarction
Time Frame: at Hospital Discharge an average of 1 day, at 1 Month, at 1 Year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants
  Hospital Discharge: number analyzed (Participants) | 555
  Hospital Discharge | 3
  1 Month: number analyzed (Participants) | 552
  1 Month | 4
  1 Year: number analyzed (Participants) | 531
  1 Year | 9

4. Secondary Outcome: Target Lesion Revascularization (TLR)
Time Frame: at Hospital Discharge an average of 1 day, at 1 Month, at 1 Year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants
  Hospital Discharge: number analyzed (Participants) | 555
  Hospital Discharge | 2
  1 Month: number analyzed (Participants) | 552
  1 Month | 3
  1 Year: number analyzed (Participants) | 531
  1 Year | 8

5. Secondary Outcome: Target Vessel Revascularization (TVR)
Time Frame: at Hospital Discharge an average of 1 day, at 1 Month, at 1 Year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants
  Hospital Discharge: number analyzed (Participants) | 555
  Hospital Discharge | 2
  1 Month: number analyzed (Participants) | 552
  1 Month | 3
  1 Year: number analyzed (Participants) | 531
  1 Year | 15

6. Secondary Outcome: Cardiac Death or Protocol-defined Any-vessel MI
Time Frame: at Hospital Discharge an average of 1 day, at 1 Month, at 1 Year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants
  Hospital Discharge: number analyzed (Participants) | 555
  Hospital Discharge | 3
  1 Month: number analyzed (Participants) | 552
  1 Month | 4
  1 Year: number analyzed (Participants) | 531
  1 Year | 9

7. Secondary Outcome: Target Lesion Failure (Cardiac Death, Protocol-defined Target Vessel MI, Clinically-driven TLR)
Time Frame: at Hospital Discharge an average of 1 day, at 1 Month, at 1 Year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants
  Hospital Discharge TLF Total: number analyzed (Participants) | 555
  Hospital Discharge TLF Total | 3
  Hospital Discharge TLF Component: Cardiac Death: number analyzed (Participants) | 555
  Hospital Discharge TLF Component: Cardiac Death | 0
  Hospital Discharge TLF Component: Protocol-defined Target Vessel MI: number analyzed (Participants) | 555
  Hospital Discharge TLF Component: Protocol-defined Target Vessel MI | 3
  Hospital Discharge TLF Component: Clinically-driven TLR: number analyzed (Participants) | 555
  Hospital Discharge TLF Component: Clinically-driven TLR | 2
  1 Month TLF Total: number analyzed (Participants) | 552
  1 Month TLF Total | 4
  1 Month TLF Component: Cardiac Death: number analyzed (Participants) | 552
  1 Month TLF Component: Cardiac Death | 0
  1 Month TLF Component: Protocol-defined Target Vessel MI: number analyzed (Participants) | 552
  1 Month TLF Component: Protocol-defined Target Vessel MI | 4
  1 Month TLF Component: Clinically-driven TLR: number analyzed (Participants) | 552
  1 Month TLF Component: Clinically-driven TLR | 2
  1 Year TLF Total: number analyzed (Participants) | 531
  1 Year TLF Total | 9
  1 Year TLF Component: Cardiac Death: number analyzed (Participants) | 531
  1 Year TLF Component: Cardiac Death | 0
  1 Year TLF Component: Protocol-defined Target Vessel MI: number analyzed (Participants) | 531
  1 Year TLF Component: Protocol-defined Target Vessel MI | 7
  1 Year TLF Component: Clinically-driven TLR: number analyzed (Participants) | 531
  1 Year TLF Component: Clinically-driven TLR | 5

8. Secondary Outcome: Target Vessel Failure (Cardiac Death, Protocol-defined Target Vessel MI, Clinically-driven TVR)
Time Frame: at Hospital Discharge an average of 1 day, at 1 Month, at 1 Year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants
  Hospital Discharge TVF Total: number analyzed (Participants) | 555
  Hospital Discharge TVF Total | 3
  Hospital Discharge TVF Component: Cardiac Death: number analyzed (Participants) | 555
  Hospital Discharge TVF Component: Cardiac Death | 0
  Hospital Discharge TVF Component: Protocol-defined Target Vessel MI: number analyzed (Participants) | 555
  Hospital Discharge TVF Component: Protocol-defined Target Vessel MI | 3
  Hospital Discharge TVF Component: Clinically-driven TVR: number analyzed (Participants) | 555
  Hospital Discharge TVF Component: Clinically-driven TVR | 2
  1 Month TVF Total: number analyzed (Participants) | 552
  1 Month TVF Total | 4
  1 Month TVF Component: Cardiac Death: number analyzed (Participants) | 552
  1 Month TVF Component: Cardiac Death | 0
  1 Month TVF Component: Protocol-defined Target Vessel MI: number analyzed (Participants) | 552
  1 Month TVF Component: Protocol-defined Target Vessel MI | 4
  1 Month TVF Component: Clinically-driven TVR: number analyzed (Participants) | 552
  1 Month TVF Component: Clinically-driven TVR | 2
  1 Year TVF Total: number analyzed (Participants) | 531
  1 Year TVF Total | 14
  1 Year TVF Component: Cardiac Death: number analyzed (Participants) | 531
  1 Year TVF Component: Cardiac Death | 0
  1 Year TVF Component: Protocol-defined Target Vessel MI: number analyzed (Participants) | 531
  1 Year TVF Component: Protocol-defined Target Vessel MI | 7
  1 Year TVF Component: Clinically-driven TVR: number analyzed (Participants) | 531
  1 Year TVF Component: Clinically-driven TVR | 12

9. Secondary Outcome: MACE (Death, Protocol-defined Any Vessel Q Wave or Non-Q Wave MI, Clinically-driven TLR
Time Frame: at Hospital Discharge an average of 1 day, at 1 Month, at 1 Year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants
  Hospital Discharge MACE Total | 4
  Hospital Discharge MACE Component: Death | 1
  Hospital Discharge MACE Component: Protocol-defined Any-Vessel Q Wave or Non-Q Wave MI: number analyzed (Participants) | 555
  Hospital Discharge MACE Component: Protocol-defined Any-Vessel Q Wave or Non-Q Wave MI | 3
  Hospital Discharge MACE Component: Clinically-driven TLR: number analyzed (Participants) | 555
  Hospital Discharge MACE Component: Clinically-driven TLR | 2
  1 Month MACE Total: number analyzed (Participants) | 554
  1 Month MACE Total | 6
  1 Month MACE Component: Death: number analyzed (Participants) | 554
  1 Month MACE Component: Death | 2
  1 Month MACE Component: Protocol-defined Any-Vessel Q Wave or Non-Q Wave MI: number analyzed (Participants) | 552
  1 Month MACE Component: Protocol-defined Any-Vessel Q Wave or Non-Q Wave MI | 4
  1 Month MACE Component: Clinically-driven TLR: number analyzed (Participants) | 552
  1 Month MACE Component: Clinically-driven TLR | 2
  1 Year MACE Total: number analyzed (Participants) | 536
  1 Year MACE Total | 17
  1 Year MACE Component: Death: number analyzed (Participants) | 536
  1 Year MACE Component: Death | 6
  1 Year MACE Component: Protocol-defined Any-Vessel Q Wave or Non-Q Wave MI: number analyzed (Participants) | 531
  1 Year MACE Component: Protocol-defined Any-Vessel Q Wave or Non-Q Wave MI | 9
  1 Year MACE Component: Clinically-driven TLR: number analyzed (Participants) | 531
  1 Year MACE Component: Clinically-driven TLR | 5

10. Secondary Outcome: Stent Thrombosis
Time Frame: at 24 Hours, at 1 Month, at 1 Year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants
  Any ARC-2 Stent Thrombosis Acute (<=24 hours) | 1
  Any ARC-2 Stent Thrombosis Sub-acute (>24 hours and <=30 days): number analyzed (Participants) | 551
  Any ARC-2 Stent Thrombosis Sub-acute (>24 hours and <=30 days) | 0
  Any ARC-2 Stent Thrombosis Late (>30 days and <=1 year): number analyzed (Participants) | 531
  Any ARC-2 Stent Thrombosis Late (>30 days and <=1 year) | 1
  Definite ARC-2 Stent Thrombosis Acute (<=24 hours) | 1
  Definite ARC-2 Stent Thrombosis Sub-acute (>24 hours and <=30 days): number analyzed (Participants) | 551
  Definite ARC-2 Stent Thrombosis Sub-acute (>24 hours and <=30 days) | 0
  Definite ARC-2 Stent Thrombosis Late (>30 days and <=1 year): number analyzed (Participants) | 531
  Definite ARC-2 Stent Thrombosis Late (>30 days and <=1 year) | 1
  Probable ARC-2 Stent Thrombosis Acute (<=24 hours) | 0
  Probable ARC-2 Stent Thrombosis Sub-acute (>24 hours and <=30 days): number analyzed (Participants) | 551
  Probable ARC-2 Stent Thrombosis Sub-acute (>24 hours and <=30 days) | 0
  Probable ARC-2 Stent Thrombosis Late (>30 days and <=1 year): number analyzed (Participants) | 531
  Probable ARC-2 Stent Thrombosis Late (>30 days and <=1 year) | 0

11. Secondary Outcome: Number of Lesions With Device Success
Description: Defined as attainment of < 30% residual stenosis of the target lesion using the assigned study stent only.
Time Frame: at Hospital Discharge an average of 1 day
Population: Device Success per lesion. Lesions that were not treated and lesions missing both site-reported and core lab-assessed percent residual stenosis were excluded from the analysis.
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Number analyzed (Lesions) | 690
Lesions | 689

12. Secondary Outcome: Number of Lesions With Lesion Success
Description: Defined as attainment of < 30% residual stenosis of the target lesion using any percutaneous method.
Time Frame: at Hospital Discharge an average of 1 day
Population: Lesion Success per lesion. Lesions that were not treated and lesions missing both site-reported and core lab-assessed percent residual stenosis were excluded from the analysis.
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Number analyzed (Lesions) | 690
Lesions | 689

13. Secondary Outcome: Number of Participants With Procedure Success
Description: Defined as attainment of < 30% residual stenosis of the target lesion using the assigned study stent only without occurrence of in-hospital major adverse cardiac events (MACE; composite of all-cause death, Q-wave or non-Q-wave MI, and any clinically-driven TLR).
Time Frame: at Hospital Discharge an average of 1 day
Population: Procedure success was analyzed per subject: for a subject to be considered a procedure success, all of the subject's target lesions had to be considered device success. Lesions that were not treated and lesions missing both site-reported and core lab-assessed percent residual stenosis were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Orsiro Sirolimus Coronary Stent System
Number analyzed (Participants) | 556
Participants | 551

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Orsiro Sirolimus Coronary Stent System
All-Cause Mortality (participants affected / at risk) | 6/556
Serious Adverse Events (participants affected / at risk) | 154/556
Other Adverse Events (participants affected / at risk) | 58/556
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orsiro Sirolimus Coronary Stent System (N=556)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 7 (7)
Angina pectoris (Cardiac disorders) | 5 (5)
Angina unstable (Cardiac disorders) | 6 (6)
Anginal equivalent (Cardiac disorders) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Arrhythmia ventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 8 (10)
Atrial flutter (Cardiac disorders) | 2 (2)
Bioprosthetic valvular thrombus (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 6 (6)
Complete heart block (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3)
Coronary artery dissection (Cardiac disorders) | 5 (5)
Coronary artery restenosis (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 17 (22)
Coronary artery thrombosis (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Oesophageal motility disorder (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Alcohol withdrawal (General disorders) | 1 (1)
Altered mental status (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 3 (3)
Catheter site haemorrhage (General disorders) | 1 (1)
Chest pain (General disorders) | 24 (25)
Non-cardiac chest pain (General disorders) | 3 (3)
Vascular stent restenosis (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Elevated liver enzyme levels (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Hepatoma (Hepatobiliary disorders) | 1 (1)
Liver mass (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 7 (7)
Cellulitis (Infections and infestations) | 2 (2)
Joint infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (6)
Pyelonephritis (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (9)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Metastatic carcinoid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered state of conciousness (Nervous system disorders) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Myasthenia gravis crisis (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Vasovegal episode (Nervous system disorders) | 1 (1)
Delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (5)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Erosion of implanted urethral mesh (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Volume depletion (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diaphragm paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Posterior pharyngeal wall hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Implantable defibrillator replacement (Surgical and medical procedures) | 1 (1)
Thymectomy (Surgical and medical procedures) | 1 (1)
Aortic aneurysm Type II endoleak (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 5 (5)
Arterial intramural haematoma (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 1 (1)
Steal syndrome (Vascular disorders) | 2 (2)
Subclavian artery stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orsiro Sirolimus Coronary Stent System (N=556)
Catheter site haematoma (General disorders) | 8 (8)
Chest pain (General disorders) | 16 (24)
Myocardial necrosis marker increased (Investigations) | 34 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT04175626/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT04175626/SAP_001.pdf